CLINICAL TRIAL: NCT01159665
Title: An Open-Label, Ascending-Exposure-Time, Single Center Trial to Evaluate the Pharmacokinetic Properties of Ocriplasmin (Generic Name of the Molecule Microplasmin) Intravitreal Injection in Subjects Scheduled for Primary Pars Plana Vitrectomy
Brief Title: The Purpose of This Study is to Evaluate the Pharmacokinetic Properties of Intravitreal Ocriplasmin Prior to Planned Primary Pars Plana Vitrectomy (PPV)
Acronym: MIVI-10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-MV-010
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-04

CONDITIONS: Vitrectomy
MeSH Terms: interventions — microplasmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- PPV 5-30 minutes after injection (Experimental): Primary Pars Plana Vitrectomy 5 to 30 minutes after 125µg of ocriplasmin intravitreal injection
  Interventions: Drug: ocriplasmin
- PPV 31-60 minutes after injection (Experimental): Primary Pars Plana Vitrectomy 31 to 60 minutes after 125µg of ocriplasmin intravitreal injection
  Interventions: Drug: ocriplasmin
- PPV 2-4 hours after injection (Experimental): Primary Pars Plana Vitrectomy 2 to 4 hours after 125µg of ocriplasmin intravitreal injection
  Interventions: Drug: ocriplasmin
- PPV 24 hours (+2 hours) after injection (Experimental): Primary Pars Plana Vitrectomy 24 hours (+2 hours)after 125µg of ocriplasmin intravitreal injection
  Interventions: Drug: ocriplasmin
- PPV 7 days (+1 day) after injection (Experimental): Primary Pars Plana Vitrectomy 7 days (+1 day)after 125µg of ocriplasmin intravitreal injection
  Interventions: Drug: ocriplasmin
- PPV without injection (No Intervention): Control Arm, no ocriplasmin intravitreal injection

INTERVENTIONS:
Drug: ocriplasmin — 125µg ocriplasmin intravitreal injection
  Other Names: microplasmin
  Arms: PPV 5-30 minutes after injection
Drug: ocriplasmin — 125µg ocriplasmin intravitreal injection
  Other Names: microplasmin
  Arms: PPV 31-60 minutes after injection
Drug: ocriplasmin — 125µg ocriplasmin intravitreal injection
  Other Names: microplasmin
  Arms: PPV 2-4 hours after injection
Drug: ocriplasmin — 125µg ocriplasmin intravitreal injection
  Other Names: microplasmin
  Arms: PPV 24 hours (+2 hours) after injection
Drug: ocriplasmin — 125µg ocriplasmin intravitreal injection
  Other Names: microplasmin
  Arms: PPV 7 days (+1 day) after injection

SUMMARY:
To evaluate the pharmacokinetic properties of intravitreal ocriplasmin 125 µg dose when administered at different time-points prior to planned primary pars plana vitrectomy (PPV)

DETAILED DESCRIPTION:
Open-label, ascending-exposure-time, single center trial in which a total of 36 subjects will be enrolled. The time to remove the vitreous will be recorded and a vitreous sample will be obtained at the beginning of vitrectomy for determination of ocriplasmin activity; 32 subjects will receive 125 μg ocriplasmin intravitreal injection prior to vitrectomy and 4 subjects will not receive ocriplasmin intravitreal injection prior to vitrectomy (control arm).

Study drug will be administered in the mid-vitreous by injection. The study eye will be examined after study drug injection to exclude retinal non-perfusion or other complications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18
* Eye disease for which a primary vitrectomy is indicated
* Best Corrected Visual Acuity (BCVA) of 20/800 or better in the non-study eye
* Written informed consent obtained from the subject prior to inclusion in the trial

Exclusion Criteria:

* Proliferative diabetic retinopathy.
* Subjects with any vitreous hemorrhage or any other vitreous opacification which precludes either of the following: visualization of the posterior pole by visual inspection OR adequate assessment of the macula by either Optical Coherence Tomography (OCT) and/or fluorescein angiogram in the study eye
* Aphakia in the study eye
* High myopia (more than 8D) in study eye (unless prior cataract extraction or refractive surgery that makes refraction assessment unreliable for myopia severity approximation, in which case axial length >28 mm is an exclusion).
* Subjects with history of rhegmatogenous retinal detachment in the either eye
* Subjects who have had ocular surgery, laser photocoagulation treatment, or intravitreal injection(s) in the study eye in the prior three months
* Subjects who have had laser photocoagulation to the macula in the study eye at any time
* Subjects with uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 26 mm Hg in spite of treatment with anti-glaucoma medication)
* Subjects with a history of uveitis in either eye.
* Subjects who are pregnant or of child-bearing potential not utilizing an acceptable form of contraception. Acceptable methods of birth control include intrauterine device, oral, implanted, or injected contraceptives, and barrier methods with spermicide.
* Subjects who, in the Investigators view, will not complete all visits and investigations
* Subjects who have participated in an investigational drug trial within the past 30 days
* Subjects who have previously participated in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Stalmans P, Girach A. Vitreous levels of active ocriplasmin following intravitreal injection: results of an ascending exposure trial. Invest Ophthalmol Vis Sci. 2013 Oct 9;54(10):6620-7. doi: 10.1167/iovs.13-11811. PMID 23982845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enroled on 15 Jul 2010 and the last patient completed the study opn 30 Nov 2010.
Pre-assignment Details: 38 subjects were enrolled into the study. However, the vitreous samples for 2 subjects were excluded from the analysis:
  * The vitreous sample for Subject 101106 was contaminated during vitrectomy.
  * Subject 101202 (Group 2) had a previous vitrectomy and retinal detachment in the study eye (exclusion criteria violation).
Groups:
- PPV 5-30 Minutes After Injection: Primary Pars Plana Vitrectomy 5 to 30 minutes after 125ug of ocriplasmin intravitreal injection
- PPV 31-60 Minutes After Injection: Primary Pars Plana Vitrectomy 31 to 60 minutes after 125ug of ocriplasmin intravitreal injection
- PPV 2-4 Hours After Injection: Primary Pars Plana Vitrectomy 2 to 4 hours after 125ug of ocriplasmin intravitreal injection
- PPV 24 Hours (+2 Hours) After Injection: Primary Pars Plana Vitrectomy 24 hours (+2 hours)after 125ug of ocriplasmin intravitreal injection
- PPV 7 Days (+1 Day) After Injection: Primary Pars Plana Vitrectomy 7 days (+1 day)after 125ug of ocriplasmin intravitreal injection
Period: Overall Study
Arm/Group | PPV 5-30 Minutes After Injection | PPV 31-60 Minutes After Injection | PPV 2-4 Hours After Injection | PPV 24 Hours (+2 Hours) After Injection | PPV 7 Days (+1 Day) After Injection | PPV Without Injection
Started | 9 | 9 | 8 | 4 | 4 | 4
Completed | 9 | 8 | 8 | 4 | 4 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PPV 5-30 Minutes After Injection | PPV 31-60 Minutes After Injection | PPV 2-4 Hours After Injection | PPV 24 Hours (+2 Hours) After Injection | PPV 7 Days (+1 Day) After Injection | PPV Without Injection | Total
Number analyzed (Participants) | 9 | 9 | 8 | 4 | 4 | 4 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (8.56) | 65.6 (13.50) | 63.8 (9.38) | 62.5 (8.66) | 59.3 (11.87) | 69.8 (7.80) | 66.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 3 | 1 | 3 | 26
  Male | 2 | 3 | 2 | 1 | 3 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Ocriplasmin Activity Levels in Vitreous Samples Obtained at the Beginning of Vitrectomy.
Description: Vitreous samples were obtained at the beginning of vitrectomy in subjects at various times relative to ocriplasmin injection (post-injection), for the determination of ocriplasmin activity (Group 1 [5-30 minutes]; Group 2 [31-60 minutes]; Group 3 [2-4 hours]; Group 4 [24 hours ±2 hours]; Group 5 [7 days ±1 day]. Subjects in Group 6 (control) did not receive the ocriplasmin injection.
Time Frame: 5-30 minutes, 31-60 minutes, 2-4 hours, 1 day, or 7 days after ocriplasmin injection
Population: Safety Set. Values for the PPV 7 days (+1 day) after injection and for PPV without injection treatment groups were all < Lower Limit of Quantification (LLOQ)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PPV 5-30 Minutes After Injection | PPV 31-60 Minutes After Injection | PPV 2-4 Hours After Injection | PPV 24 Hours (+2 Hours) After Injection | PPV 7 Days (+1 Day) After Injection | PPV Without Injection
Number analyzed (Participants) | 8 | 8 | 8 | 4 | 4 | 4
ng/mL | 11597.711 (7637.4103) | 8108.726 (5181.8506) | 2610.563 (1608.2660) | 496.473 (288.2498) | 272.370 (0.00) | 272.370 (0.00)

2. Other Pre Specified Outcome: Time Necessary to Remove the Vitreous From the Eye
Description: PPV was performed in all subjects. The time necessary to remove the vitreous from the eye, measured from first start of vitrectomy cutter till end of core vitrectomy phase, was calculated.
Time Frame: From first start of vitrectomy cutter till the end of core vitrectomy phase
Population: Safety Set
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | PPV 5-30 Minutes After Injection | PPV 31-60 Minutes After Injection | PPV 2-4 Hours After Injection | PPV 24 Hours (+2 Hours) After Injection | PPV 7 Days (+1 Day) After Injection | PPV Without Injection
Number analyzed (Participants) | 9 | 6 | 7 | 2 | 2 | 4
Minutes | 4.2 (3.07) | 3.7 (2.88) | 5.1 (1.86) | 4.5 (2.12) | 4.0 (1.41) | 4.8 (2.06)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from study drug administration through last subject follow-up visit (42 days (+ 3 days) post-surgery).
Description: Only treatment emergent AEs, defined as events with an onset on or after the date of study drug injection were included in the AE summaries. For the control arm (Group 6), AEs on or after the Baseline visit were considered treatment emergent in order to compare with the treatment groups.
Arm/Group | PPV 5-30 Minutes After Injection | PPV 31-60 Minutes After Injection | PPV 2-4 Hours After Injection | PPV 24 Hours (+2 Hours) After Injection | PPV 7 Days (+1 Day) After Injection | PPV Without Injection
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 0/8 | 0/4 | 1/4 | 2/4
Other Adverse Events (participants affected / at risk) | 2/9 | 5/9 | 5/8 | 4/4 | 4/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPV 5-30 Minutes After Injection (N=9) | PPV 31-60 Minutes After Injection (N=9) | PPV 2-4 Hours After Injection (N=8) | PPV 24 Hours (+2 Hours) After Injection (N=4) | PPV 7 Days (+1 Day) After Injection (N=4) | PPV Without Injection (N=4)
Choroidal Hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypaema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous Hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPV 5-30 Minutes After Injection (N=9) | PPV 31-60 Minutes After Injection (N=9) | PPV 2-4 Hours After Injection (N=8) | PPV 24 Hours (+2 Hours) After Injection (N=4) | PPV 7 Days (+1 Day) After Injection (N=4) | PPV Without Injection (N=4)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Chromatopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Cataract cortical (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotony of eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Metamorphosia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pupillary deformity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lens dislocation (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (2) | 2 (3) | 2 (2) | 3 (3) | 2 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dacryocistitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less